CLINICAL TRIAL: NCT01596166
Title: Efficacy of Combination Therapy With Intravenous Ketorolac and Metoclopramide for Pediatric Migraine Therapy in the Emergency Department
Brief Title: Intravenous Ketorolac and Metoclopramide for Pediatric Migraine in the Emergency Department
Acronym: EDMigraine-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDMIGR-004-01
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Probable Migraine; Migraine With Aura; Migraine Without Aura
Keywords: migraine; pediatric; childhood; emergency department; ketorolac; metoclopramide; intravenous
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders; Emergencies | interventions — Ketorolac Tromethamine; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoclopramide, Ketorolac (Experimental): 1. 10 mL/kg IV 0.9% sodium chloride
  2. Metoclopramide 0.2 mg/kg (max 10 mg) IV
  3. Ketorolac 0.5 mg/kg (max 30 mg) IV
  Interventions: Drug: Ketorolac Tromethamine; Drug: Metoclopramide
- Metoclopramide, Placebo (Placebo Comparator): 1. 10 mL/kg IV 0.9% sodium chloride
  2. Metoclopramide 0.2 mg/kg (max 10 mg) IV
  3. Placebo (normal saline)
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Ketorolac 0.5 mg/kg (max 30 mg) IV
  Other Names: Toradol; 74103-07-4
  Arms: Metoclopramide, Ketorolac
Drug: Metoclopramide — Metoclopramide 0.2 mg/kg (max 10 mg) IV
  Other Names: Maxeran; Reglan; 364-62-5

SUMMARY:
Migraine headaches are a common problem for children. When treatment at home fails, children may benefit from intravenous treatment administered in a hospital setting like the Emergency Department. Most treatments used however have only been tested in adults and the best treatment strategy for children is not always clear. The combination of more than one medication is frequently prescribed in Canadian Emergency Departments. The purpose of this study is to investigate whether the combination of ketorolac (an anti-inflammatory pain medication) and metoclopramide (an anti-nauseant that may also relieve migraine headaches) is better than metoclopramide by itself.

DETAILED DESCRIPTION:
Migraine headache is a painful condition of recurrent moderate to severe head pain associated with nausea, vomiting, photophobia, and phonophobia. The condition is highly prevalent and a significant community health problem with considerable impact on the health care system. To alleviate the pain and morbidity associated with a migraine attack, drug therapies are often employed including simple analgesics like ibuprofen and migraine-specific medications like sumatriptan. When these treatments fail or in severe, intractable cases, patients and families may present to the Emergency Department (ED).

Ketorolac in combination with metoclopramide or prochlorperazine was the most common multi-drug combination used in 36% of ED presentations for migraine across Canada in our national practice variation study. The scientific rationale for combining a non-selective non-steroidal anti-inflammatory drug (NSAID) with inhibition of both the cyclooxygenase (COX) 1 and 2 isoenzymes with other migraine therapies is enticing; however, no studies have specifically examined the relative efficacy of the practice. Why would the combination of a non-selective NSAID like ketorolac with other migraine therapies improve treatment outcomes? The benefit of multi-target combinations may be relate to the duration of the migraine and the multiple brain areas involved in sustained pain. It has long been recognized that patients who treat their migraine headaches early at the onset have a better response. The underlying mechanism for this phenomenon has now been identified. The initiation of migraine pain requires activation of the trigeminal (5th cranial nerve) nociceptive (pain) system. Activation of these sensory fibers within the arachnoid membrane on the surface of the brain produces the first and most common painful manifestation of migraine - the pulsatile headache. With each heartbeat, minor dilation of the cerebral blood vessels produces stretch and a painful activation of the trigeminal fibers known as peripheral sensitization. The second phase in the maintenance of a migraine attack over several hours is the sensitization of trigeminal pain pathways leading to higher brain centers known as central sensitization. The efficacy of medications like the triptans is greater early in the course of a migraine attack when there is only peripheral sensitization and before the onset of central sensitization. Non-selective NSAIDs like naproxen sodium and ketorolac may be uniquely effective in the reduction of central sensitization in the animal model of migraine and the reduction of migraine pain in adult patients late in the course of a migraine headache.

The population of patients in the ED is uniquely different from outpatients in that most have developed their migraine headache hours or days before presenting. In our practice variation study, the mean duration of the migraine prior to presenting to the ED was 2 days. Including an NSAID when treating a prolonged migraine in the ED may thus increase the therapeutic window and improve outcomes. While many Canadian ED physicians have adopted the practice of combining ketorolac with other migraine therapies, the gold standard assessment of efficacy and safety in a randomized clinical trial has not been applied.

ELIGIBILITY:
Inclusion Criteria:

A patient is legible to participate in this study if they meet the following criteria:

1. Patient is between 6 and 17 years of age inclusive
2. Treatment with usual therapy at home or at least one dose of oral ibuprofen or acetaminophen has not provided satisfactory relief
3. Intravenous therapy is indicated in the opinion of the treating ED physician
4. Patient has a history of migraine as defined by the International Classification of Headache Disorders - 2nd edition (Appendix 1) and meets the following criteria:

   1. During headache, at least 1 of the following: nausea and/or vomiting; two of five symptoms (photophobia, phonophobia, difficulty thinking, lightheadedness, or fatigue). Symptoms may be inferred from patient's behavior.
   2. Headache has at least 2 of the following characteristics: bifrontal/bitemporal or unilateral location; pulsating/throbbing quality; moderate or severe pain intensity; aggravation by or causing avoidance of routine physical activity. Symptoms may be inferred from patient's behavior.

Exclusion Criteria:

A patient is not eligible to participate in the study if any of the following criteria apply:

1. Patient has a contraindication to the use of metoclopramide or ketorolac in the opinion of the ED physician
2. Patient has a ventriculoperitoneal shunt
3. Patient has a fever (temperature > 38.5 oC)
4. Patient has meningismus or clinical suspicion of meningitis in the opinion of the ED physician
5. Patient has a history of head trauma causing headache in the last 1 week prior to presentation to the ED
6. Patient is unable to complete the efficacy assessments (e.g. language barrier)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mean reduction in pain intensity | 2 hours
  Measured on Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Pain freedom | 2 hours
  VAS=0
Headache relief - 33 | 2 hours
  Defined as a 33% reduction on the VAS.
Headache relief - 50 | 2 hours
  Defined as a 50% reduction on the VAS
Presence of nausea | 2 hours
Presence of vomiting | 2 hours
Use of rescue medications | 2 hours
  Permitted per protocol 60 minutes after start if intravenous infusion.
Sustained pain-free | 25 hours
  No recurrence of headache within 24 hours if pain was completely eliminated (VAS = 0) prior to discharge.
Sustained headache relief | 24 hours
  No increase in headache by 33% on the VAS or 50% on the VAS if headache relief was initially achieved.
Minimum clinically significant difference | 2 hours
  1. "I would take the medication again"
  2. "My headache is a bit better/worse"
  3. "My headache is a lot better/worse"
Adverse events | 2 hours
  All serious and non-serious adverse events including akathisia and dystonia.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Richer, MD, MSc, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta